CLINICAL TRIAL: NCT00907387
Title: A Phase 2, Double-Blind, Randomized, Parallel-Group, Controlled, Dose-Ranging, Multi-Center Study to Evaluate the Safety and Efficacy of RT001, a Botulinum Toxin Type A Topical Gel, for the Treatment Lateral Canthal Lines in Adults
Brief Title: Safety and Efficacy Study of RT001 to Treat Moderate to Severe Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL010LCL
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Lateral Canthal Lines
Keywords: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
MeSH Terms: interventions — RT001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose A (Active Comparator): Dose A RT001
  Interventions: Drug: RT001
- Dose B (Active Comparator): Dose B RT001
  Interventions: Drug: RT001
- Dose C (Placebo Comparator): Dose C Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RT001 — Dose A RT001
  Arms: Dose A
Drug: RT001 — Dose B RT001
  Arms: Dose B
Other: Placebo — Dose C Placebo
  Arms: Dose C

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of RT001 to treat moderate to severe lateral canthal lines in adults and duration of effect.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel-group, controlled, dose-ranging, multi-center study to evaluate the safety and efficacy of RT001 compared to placebo applied as a single, bilateral application in at least 180 subjects with moderate to severe LCLs. Subjects will be randomized within each site to 1 of 3 treatment groups in a 1:1:1 ratio. The safety and efficacy of two different doses of RT001, compared to placebo, will be evaluated.

At least 180 adult volunteers who have provided informed consent and have met the study eligibility criteria will be enrolled. Subjects will be enrolled in two (2) sequential cohorts. Cohort 1 will consist of 72 subjects; 24 subjects per treatment group. Cohort 2 will consist of 108 subjects; 36 subjects per treatment group. In order to confirm the safety of the test articles, Cohort 2 will not be enrolled until all Cohort 1 subjects have reached Day 14 or later with no Study Pause Criteria being observed.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 30 to 60 years of age
* Bilateral lateral canthal lines rated as moderate or severe
* Willing to refrain from receiving facial fillers, laser treatments, use of any product that affects skin remodeling or a product that may cause an active dermal response in the treatment area beginning at Screening and through End of Study
* Women of childbearing potential must be practicing and willing to continue to use an effective method of birth control during the course of the study

Exclusion Criteria:

* Muscle weakness or paralysis in the area receiving study treatment -Active skin disease or irritation at the treatment areas
* Undergone any procedures that may affect the lateral canthal region during the past 12 months prior to Screening
* Use of a topical steroid on either of the treatment areas or use of medications that suppress the immune system 30 days prior to Screening and continuing through End of Study (Day 28)
* Any abnormality on the electrocardiogram (ECG) at Screening or any history of clinically significant arrhythmia, unstable angina, myocardial infarction or congestive heart failure.
* Previous treatment with Botulinum Toxin Type A in the face area

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment at Rest from Baseline (Day 0) to Day 28 | Day 28

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Tranowski, Study Director — Revance Therapeutics, Inc.
Locations (9):
- United States (9):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Richard G. Glogau, Inc., San Francisco, California
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - SkinCare Physicians, Inc., Chestnut Hill, Massachusetts
  - Skin Specialists, PC, Omaha, Nebraska
  - Head and Neck Surgical Group, New York, New York
  - Aesthetic Plastic Surgery, New York, New York
  - Dermatology Surgery and Laser Center, White Plains, New York
  - Suzanne Bruce & Associates / The Center for Skin Research, Houston, Texas